CLINICAL TRIAL: NCT02935387
Title: REMission INDuction in Very Early Rheumatoid Arthritis
Acronym: REMINDRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Jacob M van Laar, Professor, MD PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REMINDRA
Record Dates: First submitted 2016-10-10; First posted 2016-10-17 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Very early rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taper methotrexate, then golimumab (Experimental): Taper methotrexate 25>0mg/wk during 24 weeks, then, if still in sustained remission, taper golimumab 50>0mg/month during 24 weeks.
  Interventions: Other: Taper
- Taper golimumab, then methotrexate (Active Comparator): Taper golimumab 50>0mg/month during 24 weeks, then, if still in sustained remission, taper methotrexate 25>0mg/wk during 24 weeks.
  Interventions: Other: Taper

INTERVENTIONS:
Other: Taper — Taper

SUMMARY:
Rheumatoid arthritis (RA) patients in remission with a combination of TNFinhibitors (TNFi) and methotrexate (MTX) often express their wish to stop MTX treatment because of side effects. Given the efficacy of TNFi it is conceivable that in early RA patients in remission with methotrexate (MTX)/TNFi stepwise discontinuation of MTX prior to TNFi is superior in maintaining sustained remission and reaching drug free remission as compared to discontinuation of TNFi prior to MTX.

Objective: To investigate whether tapering MTX first, then the TNFi golimumab (GOL), is more efficacious than tapering GOL first, then MTX, in sustaining remission and reaching drug free remission.

Study design: multicenter, open label clinical trial in very early RA patients. Remission will be induced by an open label treat-to-target (T2T) remission induction protocol in clinical care: (MTX, hydroxychloroquine (HCQ), i.m. glucocorticoids (GC), and, if not in remission, the TNFi golimumab (GOL)) (phase I, 3/4th or 1 year). Patients in sustained remission on MTX/GOL (DAS28<2.6 with max 4 swollen joints of the 44 swollen joint count (SJC) at 2 consecutive visits 3 months apart) will be randomized to taper either MTX first, then GOL or GOL first, then MTX with as primary endpoint sustained (drug free) remission (phase II, 1 year). During 1 year additional follow-up maintenance of drug-free sustained remission will be investigated (phase III).

Study population: RA patients fulfilling 2010 American College of Rheumatology (ACR)/EUropean League Against Rheumatism (EULAR) criteria for RA, with symptom duration <12 months; naïve for anti-rheumatic drugs and glucocorticoids for RA; DAS28 ≥3.2.

Intervention: Patients in sustained remission (defined as DAS28<2.6 with max 4 swollen joints of the 44SJC at ≥ 2 consecutive visits 3 months apart) on MTX/GOL at the end of phase I (after 24 weeks of treatment with MTX/GOL) will be randomized in a ratio of 1:1 to taper medication as follows:

* Taper and stop GOL first during 24 weeks, then, if still in sustained remission, taper and stop MTX during 24 weeks
* Taper and stop MTX first during 24 weeks, then, if still in sustained remission, taper and stop GOL during 24 weeks The primary end point is the proportion of patients in sustained remission at week 24 after start of tapering of either MTX or GOL first. The main secondary end point is the proportion of patients in drug-free sustained remission, at week 48 after start of tapering.

DETAILED DESCRIPTION:
Secondary endpoints:

Phase I (Remission induction):

* The proportion of patients on MTX/HCQ/GC in remission, defined as DAS28<2.6, at week 12 or week 24 after start of treatment.
* The proportion of patients on MTX/GOL in sustained remission, defined as DAS28<2.6 with max 4 swollen joints of the 44SJC at 2 consecutive visits 3 months apart, at week 24 after start of GOL treatment.
* Predictors of remission upon treatment with MTX, HCQ and a single injection of i.m. GC (e.g. smoking status, BMI, alcohol use, sex, disease duration, DAS28, Rheumatoid Factor (RF) -status, Anti-citrullinated protein antibody (ACPA) -status, presence of erosions)
* Predictors of remission upon treatment with MTX and GOL (e.g. smoking status, BMI, alcohol use, sex, disease duration, DAS28, RF-status, ACPA-status, presence of erosions)

Phase II (Tapering):

* The proportion of patients in sustained remission, defined as DAS28<2.6 with max 4 swollen joints of the 44SJC at 2 consecutive visits 3 months apart, at week 48 after start of tapering MTX first, then GOL or GOL first, then MTX.
* The proportion of patients in drug-free sustained remission, defined as DAS28<2.6 with max 4 swollen joints of the 44SJC at 2 consecutive visits 3 months apart while off anti-rheumatic treatment, at week 48 after start of tapering
* Mean disease activity, using the disease activity score assessing 28 joints (DAS28), at week 24 and week 48 after start of tapering
* Mean functional ability, using the Dutch consensus health assessment questionnaire (HAQ), at week 24 and week 48 after start of tapering
* Mean quality of life, using the visual analogue scale (VAS) of the EuroQol 5 dimensions (EQ5D) questionnaire, at week 24 and week 48 after start of tapering
* Mean anxiety and depression (using the Hospital Anxiety and Depression Scale (HADS)), at week 24 and week 48 after start of tapering
* Mean fatigue (using the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F)), at week 24 and week 48 after start of tapering
* The proportion of serious adverse events (SAEs) in the two tapering strategies after 24 and after 48 weeks.
* The time until remission (DAS28<2.6) after retreatment with the last effective dose upon flare while tapering MTX/GOL.

Phase III (Follow-up):

* The proportion of patients in drug-free sustained remission, defined as DAS28<2.6 with max 4 swollen joints of the 44SJC at 2 consecutive visits 3 months apart while off anti-rheumatic treatment, at week 48 after discontinuation of both MTX and GOL
* The time until remission, defined as DAS28<2.6, after retreatment in clinical care upon flare
* The proportion of serious adverse events (SAEs) in the two tapering strategies at week 24 and week 48.

Phase II and III:

* Cost per extra patient in remission up to week 96 after start of tapering (end of phase III)
* Cost per Quality Adjusted life Year (QALY) gained up to week 96 after start of tapering (end of phase III)

Overall:

- The sensitivity and predictive value of the patient reported Routine Assessment of Patient Index Data 3 (RAPID3) to detect remission and flare

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling 2010 ACR/EULAR criteria for RA.
* Patient reported symptom duration < 12 months
* Naïve for DMARD and biological treatment
* Naïve for previous use of glucocorticoids for RA
* DAS28 ≥3.2

Exclusion Criteria:

* Being pregnant or being a nursing women or a women of child bearing potential without (adequate) use of contraception
* Having any other inflammatory rheumatic disease than RA, except for secondary Sjögren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
proportion of patients in sustained remission | At week 24 after start of tapering
  the proportion of patients in sustained remission at week 24 after start of tapering of either MTX or GOL first.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M van Laar, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Reumazorg Zuidwest Nederland, Goes
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No